CLINICAL TRIAL: NCT03411668
Title: The Effectiveness of an Evidence Based Practice (EBP) Educational Programme in Undergraduate Nursing Students' EBP Beliefs and Knowledge, and the Extent of Their EBP Implementation: A Cluster Randomized Control Trial
Brief Title: EBP Educational Programme in Nursing Students' EBP Beliefs and Knowledge, and the Extent of Their EBP Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Enfermagem de Coimbra (Other)
Collaborators: University of Coimbra (Other)
Responsible Party: Principal Investigator, Daniela Cardoso, Researcher Grant Holder, Escola Superior de Enfermagem de Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EBP_Educ_Nurs
Record Dates: First submitted 2018-01-20; First posted 2018-01-26 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Evidence-Based Nursing
Keywords: undergraduate nursing students; evidence based practice beliefs; evidence based practice knowledge; evidence based practice implementation; Evidence based practice Education programme

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assignment to the arms will be made by an independent researcher using random.org.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBP Educational Programme (Experimental): The educational EBP programme will include 12 hours of classroom lessons regarding EBP more 6 hours of mentorship made to a small groups of students (2 or 3 students per group).
  Interventions: Other: EBP Educational Programme
- Usual Educational Programme (No Intervention): Without intervention. The participants in this group will be maintain usual educational programme.

INTERVENTIONS:
Other: EBP Educational Programme — The educational EBP programme will include 12 hours of classroom lessons regarding EBP more 6 hours of mentorship made to a small groups of students (2 or 3 students per group).
  Arms: EBP Educational Programme

SUMMARY:
Evidence-based practice (EBP) prevents unsafety/inefficiency and improves healthcare quality. However, EBP implementation and sustainment are challenging for healthcare organizations and providers considering gaps between research and practice. An educational preparation of the future healthcare professionals can minimize these gaps. Thus, it is mandatory that undergraduate curricula in health sciences, namely in nursing, promote an EBP culture so that future health professionals use it into clinical practice. Within the Portuguese context, there is no available scientific literature about the current state of EBP integration in the undergraduate nursing curricula. Thereby, the investigators intend to verify if an EBP educational programme would be successful in improving the undergraduate nursing students' EBP knowledge and beliefs and, and the extent of their EBP implementation This will be tested using a prospective cluster randomized control trial with two-armed parallel group design.

DETAILED DESCRIPTION:
Evidence-Based Practice (EBP), also known as Evidence-Informed Practice, could be defined as a "clinical decision-making that considers the best available evidence; the context in which the care is delivered; client preference; and the professional judgment of the health professional".

It has been recognizing that the adoption, implementation and sustainment of EBP in healthcare organizations are very important to promotes high-value health care, improves the patient experience and health outcomes, and reduces health care costs.

In consequence, several organizations acclaim EBP implementation, because this implementation improves the quality of care; reduces the uncertainty, risk and variability; and becomes the decision-making more simplified. Moreover, Dawes et al at the "Sicily statement on evidence-based practice" highlighted that "all health care professionals need to understand the principles of EBP, recognize EBP in action, implement evidence-based policies, and have a critical attitude to their own practice and to evidence".

Nevertheless, nowadays EBP is not the standard of care in the world and some studies recognized education as a strategy to promotes the adoption, implementation and sustainment of EBP.

In fact, the Committee on the Health Professions Education Summit in 2003 recommended the development of competencies regarding the EBP use in all health professional educational programs. Therefore, it is important that undergraduate nursing curricula are based on EBP principles to educate the future nurses to use EBP into clinical practice. This will, consequently, improve health outcomes, with a positive impact in patients' safety, costs and health systems. Regardless of the above recommendation, the nursing curricula still provide contents related to traditional nursing research and do not integrate the EBP content and process.

Therefore, this randomized control trial aims to evaluate the effectiveness of an educational EBP programme in undergraduate nursing students' EBP beliefs and knowledge, and the extent of their EBP implementation. This study will have two arms: experimental group (EBP educational program) and control group (no intervention - education as usual) and it will have the following methodology:

* Sample: For sample size calculation it was used the software G*Power 3.1.9.2. Power analysis was based on a type I error of 0.05; power of 0.80; effect size f=0.25; and ANOVA: repeated measures between factors determined a total sample size of 92. In a Portuguese nursing school, six optional courses of the 8th semester of the nursing graduation were randomly assigned to experimental (EBP educational programme) or control group (no intervention - education as usual). An independent researcher performed this assignment using random.org.
* Intervention: The EBP educational programme will be implemented over 17 weeks (12 hours of lessons - expositive method and practice method and 3 sessions of mentorship to small groups of students - 2/3 students - with the duration of 2 hours each).
* Assessment: All participants will be assessed before (week 0) and after the intervention (week 18) by a blind assessor using the validated instruments to assess undergraduate nursing students' EBP beliefs, the extent of their EBP implementation and their knowledge in EBP.
* Data analysis: The data will be analyzed using Statistical Package for the Social Sciences (SPSS) to conduct a descriptive and inferential analysis. To minimize the noncompliance impact, the intention to treat analysis - Last observation carried forward will be used.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students, aged 18 years or older, attending the 8th semester of the degree course in nursing at a nursing school in Portugal

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the participant's Evidence Based Practice knowledge | Post-intervention assessment (week 18)
  Outcome measure: "Fresno Test" of Ramos, Schafer, & Tracz (2003) - adapted to nursing students and Portuguese population

SECONDARY OUTCOMES:
Change from Baseline in the participant's Evidence Based Practice beliefs | Post-intervention assessment (week 18)
  Outcome measure: Evidence Based Practice beliefs scale of Melnyk, Fineout-Overholt, & Mays (2008) - Portuguese version.
  Minimum score: 16; maximum score: 80. Higher values represent a better outcome.
Change from Baseline in the participant's Evidence Based Practice implementation | Post-intervention assessment (week 18)
  Outcome measure: Evidence Based Practice implementation scale for students of Melnyk, Fineout-Overholt, & Mays (2008) - Portuguese version.
  Minimum score: 0; maximum score: 72. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Cardoso, RN, Principal Investigator — UICISA: E, ESEnfC/Faculty of Medicine, University of Coimbra
Locations (1):
- ESEnfC, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Apostolo J, Cardoso D, Rodrigues MA. It takes three to tango: embracing EBP. JBI Database System Rev Implement Rep. 2016 Apr;14(4):1-2. doi: 10.11124/JBISRIR-2016-2889. No abstract available. PMID 27532303
- [Background] Asokan GV. Evidence-based practice curriculum in allied health professions for teaching-research-practice nexus. J Evid Based Med. 2012 Nov;5(4):226-31. doi: 10.1111/jebm.12000. PMID 23557503
- [Background] Black AT, Balneaves LG, Garossino C, Puyat JH, Qian H. Promoting evidence-based practice through a research training program for point-of-care clinicians. J Nurs Adm. 2015 Jan;45(1):14-20. doi: 10.1097/NNA.0000000000000151. PMID 25390076
- [Background] Institute of Medicine (US) Committee on the Health Professions Education Summit; Greiner AC, Knebel E, editors. Health Professions Education: A Bridge to Quality. Washington (DC): National Academies Press (US); 2003. Available from http://www.ncbi.nlm.nih.gov/books/NBK221528/ PMID 25057657
- [Background] Dawes M, Summerskill W, Glasziou P, Cartabellotta A, Martin J, Hopayian K, Porzsolt F, Burls A, Osborne J; Second International Conference of Evidence-Based Health Care Teachers and Developers. Sicily statement on evidence-based practice. BMC Med Educ. 2005 Jan 5;5(1):1. doi: 10.1186/1472-6920-5-1. PMID 15634359
- [Background] Mazurek Melnyk B, Newhouse R. Evidence-based practice versus evidence-informed practice: a debate that could stall forward momentum in improving healthcare quality, safety, patient outcomes, and costs. Worldviews Evid Based Nurs. 2014 Dec;11(6):347-9. doi: 10.1111/wvn.12070. Epub 2014 Nov 13. No abstract available. PMID 25394811
- [Background] Melnyk BM, Fineout-Overholt E, Mays MZ. The evidence-based practice beliefs and implementation scales: psychometric properties of two new instruments. Worldviews Evid Based Nurs. 2008;5(4):208-16. doi: 10.1111/j.1741-6787.2008.00126.x. PMID 19076922
- [Background] Melnyk BM, Fineout-Overholt E, Gallagher-Ford L, Kaplan L. The state of evidence-based practice in US nurses: critical implications for nurse leaders and educators. J Nurs Adm. 2012 Sep;42(9):410-7. doi: 10.1097/NNA.0b013e3182664e0a. PMID 22922750
- [Background] Melnyk BM, Gallagher-Ford L, Long LE, Fineout-Overholt E. The establishment of evidence-based practice competencies for practicing registered nurses and advanced practice nurses in real-world clinical settings: proficiencies to improve healthcare quality, reliability, patient outcomes, and costs. Worldviews Evid Based Nurs. 2014 Feb;11(1):5-15. doi: 10.1111/wvn.12021. Epub 2014 Jan 21. PMID 24447399
- [Background] Oh EG, Kim S, Kim SS, Kim S, Cho EY, Yoo JS, Kim HS, Lee JH, You MA, Lee H. Integrating evidence-based practice into RN-to-BSN clinical nursing education. J Nurs Educ. 2010 Jul;49(7):387-92. doi: 10.3928/01484834-20100331-02. Epub 2010 Mar 31. PMID 20411864
- [Background] Ramos KD, Schafer S, Tracz SM. Validation of the Fresno test of competence in evidence based medicine. BMJ. 2003 Feb 8;326(7384):319-21. doi: 10.1136/bmj.326.7384.319. PMID 12574047
- [Background] Directorate-General of Health, Ministry of Health. (2012). National Health Plan 2012-2016. Lisbon, Portugal: author. Retrieved from http://pns.dgs.pt/pns-versao-completa/
- [Background] International Council of Nurses. (2012). Closing the Gap: from Evidence to Action. Geneva: author. ISBN: 978-92-95094-75-8
- [Background] Ordem dos Enfermeiros. (2006). Tomada de Posição sobre Investigação em Enfermagem. Lisboa: author. Retrieved from http://www.ordemenfermeiros.pt/tomadasposicao/Documents/TomadaPosicao_26Abr2006.pdf
- [Background] Mohsen, M. M., Safaan, N. A., & Okby, O. M. (2016). Nurses' Perceptions and Barriers for Adoption of Evidence Based Practice in Primary Care: Bridging the Gap. American Journal of Nursing Research, 4(2), 25-33.
- [Background] Pearson A, Wiechula R, Court A, Lockwood C. The JBI model of evidence-based healthcare. Int J Evid Based Healthc. 2005 Sep;3(8):207-15. doi: 10.1111/j.1479-6988.2005.00026.x. PMID 21631749